CLINICAL TRIAL: NCT03415412
Title: Clinical Evaluation of Three Different Universal Adhesives and a Universal Flowable Composite for Restoration of Non-carious Cervical Lesions
Brief Title: Clinical Evaluation of Three Different Universal Adhesives in Non-carious Cervical Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCCLsclinic
Record Dates: First submitted 2017-12-23; First posted 2018-01-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Tooth Diseases
Keywords: non-caries cervical lesion; universal adhesives
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group CU (Clearfil Universal) (Experimental): Clearfil Univesal Bond (Kuraray Dental, New York, United States of America), adhesive system
  Interventions: Device: Clearfil Univesal Bond
- Group IU (Ibond Universal) (Experimental): IBond Universal (Heraeus Kulzer GmbH, Hanau, Germany), adhesive system
  Interventions: Device: IBond Universal
- Group GP (G-Premio) (Experimental): G-Premio Bond (GC Coorporation, Tokyo, Japan), adhesive system
  Interventions: Device: G-Premio Bond

INTERVENTIONS:
Device: Clearfil Univesal Bond — Adhesive systems
  Arms: Group CU (Clearfil Universal)
Device: IBond Universal — Adhesive systems
  Arms: Group IU (Ibond Universal)
Device: G-Premio Bond — Adhesive systems
  Arms: Group GP (G-Premio)

SUMMARY:
The aim of this randomized, controlled prospective clinical trial is to evaluate and compare the performances of three different universal adhesives using a flowable universal composite resin in the restoration of non-caries cervical lesions over 48-month period.Participants over 18 will be included to the study. Oral hygiene instructions will be given before procedures. All the lesions will be restored by the same clinician who will not participate to the selection of patients for eligibility. Each patient will receive at least three restorations and randomization will be applied using a table of random numbers. All lesions will be cleaned before restoring. Adhesive procedures and restorations will be placed according to manufacturers' recommandation.

The flowable universal composite resin will be placed in bulk and light-cured for 40 seconds. The restorations will be contoured and polished with Optidisc discs (Kerr Coorporation, Orange, CA, USA).

Patients will be recalled at baseline and will be recalled at control periods after placement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old with 20 teeth under occlusion. They will be required to have at least three NCCLs needed restoration in different teeth. All the NCCLs selected were in similar sizes varying between 1-3 mm.

Exclusion Criteria:

* Patients with severe periodontal disease, rampant, uncontrolled caries, xerostomia, serious medical problems preventing them from attending review visits, poor gingival health, heavy bruxism and removable partial dentures will not be included in the present study. Also, participiants will be excluded, if they are undergoing bleaching treatment or orthodontic treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different universal adhesives | Two years
  Two year results according to USPHS criteria

REFERENCES:
- [Derived] Oz FD, Ozturk C, Soleimani R, Gurgan S. Sixty-month follow up of three different universal adhesives used with a highly-filled flowable resin composite in the restoration of non-carious cervical lesion. Clin Oral Investig. 2022 Aug;26(8):5377-5387. doi: 10.1007/s00784-022-04505-x. Epub 2022 Apr 27. PMID 35477817